CLINICAL TRIAL: NCT07309445
Title: A Multicenter, Prospective, Longitudinal Study to Assess Real-World Use and Outcomes After the Launch of TAR-200 for NMIBC in the US
Brief Title: A Study to Assess Real-World Use and Outcomes of TAR-200 for Participants With Non-Muscle Invasive Bladder Cancer (NMIBC) in the United States
Acronym: Nova-sTAR
Status: Not yet recruiting | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 17000139BLC4004; 17000139BLC4004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Non-Muscle Invasive Bladder Neoplasms
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NMIBC Participants: Routine Clinical Practice Setting: Participants with confirmed diagnosis of NMIBC and who have initiated first dose of TAR-200 in a real-world clinical setting, within 6 weeks prior to baseline visit/Study visit 1 will be observed for 24 months from the initiation of the first dose of TAR-200, or until the participant dies, is lost to follow-up, or withdraws consent in the study. No intervention will be administered as a part of this study.

SUMMARY:
The purpose of this study is to assess how well TAR-200 works in real-word by measuring the time taken from the first TAR-200 insertion to worsening of cancer or until the signs and symptoms of cancer occur again (disease-free survival) in participants with non-muscle invasive bladder cancer (NMIBC; an early-stage bladder cancer that is limited to the inner lining of bladder).

ELIGIBILITY:
Inclusion criteria:

* Has a confirmed diagnosis of NMIBC based on TURBT or cold cup biopsy
* Initiated first dose of TAR-200 in a real-world setting within 6 weeks prior to baseline visit/Study visit 1
* Participants with childbearing potential are required to adhere to contraceptive recommendations as specified in the approved product labeling for TAR-200. Additionally, participants should seek consultation with their physician for personalized contraceptive advice
* Must provide informed consent as described in the protocol

Exclusion criteria:

* Has any medical condition deemed by the health care practitioner (HCP) as contraindicated to receive TAR-200 treatment
* Had previous treatment with TAR-200 discontinued prior to baseline visit/Study visit 1
* Previously received TAR-200 intravesically as part of a clinical trial(s)
* Previously received greater than (>) 2 doses/cycles of TAR-200 in the real-world setting
* Currently participating in an interventional bladder cancer clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants aged 18 years or above with confirmed diagnosis of NMIBC (based on transurethral resection of bladder tumor [TURBT] or cold cup biopsy), who initiated the first dose of TAR-200 in a real-world setting within 6 weeks prior to baseline visit/Study visit 1 and willing to provide informed consent will be enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-12-18 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | Up to 24 months
  DFS is defined as the time from first TAR-200 initiation date to the time of the first recurrence of NMIBC (Ta, any T1 or carcinoma in-situ [CIS)], progression (to muscle invasive bladder cancer [MIBC; T greater than or equal to {>=} 2] or to lymph node [N+] or to distant disease [M+], whichever occurs first), or death due NMIBC, whichever occurs first.

SECONDARY OUTCOMES:
Complete Response (CR) Rate | At 3, 6, 12, 18, and 24 months
  CR rate is defined as the percentage of participants achieving a CR at any time after the initial TAR-200 treatment. CR is defined as the total absence of NMIBC (both CIS and papillary) per investigator assessment.
Duration of Response (DOR) | Up to 24 months
  DOR is defined as the interval between the noted date of first complete response of any kind to TAR-200 and the date on which recurrence of NMIBC (Ta, any T1 or CIS), progressive disease or death due to NMIBC occurs, whichever occurs first.
Overall Survival (OS) | Up to 24 months
  OS is defined as the interval between the date of the first TAR-200 administration and date of death due to any cause.
Cancer-Specific Survival (CSS) | Up to 24 months
  CSS is defined as the interval between the date of the first TAR-200 insertion and date of death due to bladder cancer or if cause of death is unknown.
Time to Next Treatment (TTNT) | Up to 24 months
  TTNT is defined as the time difference from the first TAR-200 insertion date to the start date of next bladder cancer treatment.
Number of Participants with Radical Cystectomy (RC) /Bladder-Intact Survival | Up to 24 months
  Radical cystectomy or bladder-intact survival is defined as the time from first TAR-200 insertion date to the date of the first evidence of radical cystectomy.
Time to RC /Bladder-Intact Survival | Up to 24 months
  Radical cystectomy or bladder-intact survival is defined as the time from first TAR-200 insertion date to the date of the first evidence of radical cystectomy.
Number of Participants with Adverse Events (AEs) | Up to 24 months
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the treatment. Severity of AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0. by using standard grades as follows: Grade 1: Mild; asymptomatic or mild symptoms; Grade 2: Moderate; minimal, local or noninvasive intervention indicated; Grade 3: Severe but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; Grade 4: Life-threatening consequences; and Grade 5: Death related to AE. AE related to TAR-200 treatment and/or TAR-200 procedure (that is, insertion and removal of TAR-200 or its urinary placement catheter [UPC]) will be reported.
Treatment Patterns for TAR-200 | Up to 24 months
  Treatment patterns, including frequency, adherence, sequencing, and reasons for initiation, interruption, and discontinuation of treatment, and subsequent line of treatment (including re-treatment with TAR-200) will be reported.
Time to TAR-200 Discontinuation | Up to 24 months
  Time to TAR-200 discontinuation will be reported.
Study Dropout Rate | Up to 24 months
  Study dropout rate and reason for dropout from the study will be reported.
Treatment Adherence: Impact of Follow-up Reminders | Up to 24 months
  Number of participants who adhered to treatment after follow-up reminders will be reported.
DFS After Re-Treatment with TAR-200 | Up to 24 months
  Re-treatment is defined as treating a participant with TAR-200 after NMIBC recurrence and may follow Transurethral Resection of bladder tumor (TURBT) for papillary disease or cold cup biopsy for CIS only recurrence. DFS is defined as the time from first TAR-200 initiation date to the time of the first recurrence of NMIBC (Ta, any T1 or CIS), progression (to MIBC [T greater than or equal to {>=} 2] or to lymph node [N+] or to distant disease [M+], whichever occurs first), or death due to NMIBC, whichever occurs first.
CR Rate After Re-treatment with TAR-200 | Up to 24 months
  Re-treatment is defined as treating a participant with TAR-200 after NMIBC recurrence and may follow TURBT for papillary disease or cold cup biopsy for carcinoma in-situ (CIS) only recurrence. CR rate is defined as the percentage of participants achieving a CR at any time after the TAR-200 re-treatment. CR is defined as the total absence of NMIBC (both carcinoma in-situ [CIS] and papillary) per investigator assessment.
DOR After Re-Treatment with TAR-200 | Up to 24 months
  Re-treatment is defined as treating a participant with TAR-200 after NMIBC recurrence and may follow TURBT for papillary disease or cold cup biopsy for CIS only recurrence. DOR is defined as the interval between the noted date of first complete response of any kind to TAR-200 and the date on which recurrence of NMIBC (Ta, any T1 or CIS), progressive disease or death due to NMIBC occurs, whichever occurs first.
OS After Re-Treatment with TAR-200 | Up to 24 months
  Re-treatment is defined as treating a participant with TAR-200 after NMIBC recurrence and may follow TURBT for papillary disease or cold cup biopsy for CIS only recurrence. OS is defined as the interval between the date of the first TAR-200 re-administration and date of death due to any cause.
CSS After Re-Treatment with TAR-200 | Up to 24 months
  Re-treatment is defined as treating a participant with TAR-200 after NMIBC recurrence and may follow TURBT for papillary disease or cold cup biopsy for CIS only recurrence. CSS is defined as the interval between the date of the TAR-200 re-insertion and date of death due to bladder cancer or if cause of death is unknown.
TTNT After Re-Treatment with TAR-200 | Up to 24 months
  Re-treatment is defined as treating a participant with TAR-200 after NMIBC recurrence and may follow TURBT for papillary disease or cold cup biopsy for CIS only recurrence. TTNT is defined as the time difference from TAR-200 re-insertion date to the start date of next bladder cancer treatment.
Number of Participants with Radical cystectomy/ Bladder-Intact Survival After Re-Treatment with TAR-200 | Up to 24 months
  Re-treatment is defined as treating a participant with TAR-200 after NMIBC recurrence and may follow TURBT for papillary disease or cold cup biopsy for CIS only recurrence. Radical cystectomy or bladder-intact survival is defined as the time from TAR-200 re-insertion date to the date of the first evidence of radical cystectomy.
Time to RC /Bladder-Intact Survival After Re-Treatment with TAR-200 | Up to 24 months
  Re-treatment is defined as treating a participant with TAR-200 after NMIBC recurrence and may follow TURBT for papillary disease or cold cup biopsy for CIS only recurrence. Radical cystectomy or bladder-intact survival is defined as the time from TAR-200 re-insertion date to the date of the first evidence of radical cystectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency